CLINICAL TRIAL: NCT04034303
Title: Natural History, Risk Factors and Predictive Biomarkers for Celiac Disease: a Prospective Multicenter Study.
Brief Title: Risk Factors for the Development of Celiac Disease in Genetically Predisposed Children
Acronym: NEOCEL
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Renata Auricchio, Dr., Federico II University
Other Study IDs: NEOCEL2019
Record Dates: First submitted 2019-07-24; First posted 2019-07-26 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: Prevention of Clinical Symptoms in Celiac Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples for serum, cells, nucleic acids Urine for metabolomic Analysis Breast Milk for metabolomic analysis Feces for microbiome
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: analysis of genetic and epigenetic risk factors — analysis of gene, methylation and expression, microbiome

SUMMARY:
The study aims to identify risk factors for the development of Celiac Diseases in families with a recognized genetic risk for the presence of a confirmed proband case. Candidate mother will be recruited before a planned pregnancy or within the first 12 weeks of pregnancy. Familial and environmental risk factors will be evaluated within the couple of parents. Pregnancy will be followed up and appropriate biological samples collected. Delivery will be supervised in order to collect biological samples. Newborns will be controlled from birth up to the 6th year of age. Data about clinical events related to health, life attitudes, nutrition will be collected together with biological samples either in the pregnant mother as well as in the infant.

DETAILED DESCRIPTION:
* CD epidemics: Celiac Disease incidence is increasing at unexpected rates in the last two decades in all gluten-consuming populations.
* Remarkable stratified genetic risk: there is a strong genetic component as the main risk to develop disease, as supported by > 85% concordance in monozygotic twins, but genetics cannot change over decades and does not explain the epidemic which has been observed. The presence of double HLA DQ2 in female subjects does increases the risk of disease above that of a mendelian recessive inheritance. Hence the estimation of environmental factors associated to the genetic risk is quite complex and does need a very strict prospective longitudinal study design, since each factor is likely to produce, if ever, a quite small odds ratio .
* Gene expression in the first year of life: we have observed, in our previous cohort studies, that the expression of at least a small set of CD associated candidate genes is substantially different between the children who eventually develop Cd and those who do not, already a 6 months of age, much before any measurable recognition of the gluten antigen, development of antibodies or any clinical sign (ref 3 Galatola).
* Epigenetic changes in small intestinal tissue: in addition of the previously reported gene expression differences, gene methylation and related expression of CD associated candidate genes have been observed in the epithelium and the lamina propria of Cd patients . In addition, microRNA appear to be differently expressed in patients versus controls.
* Early events in the first-second year of life before diagnosis: our groups and others observed that the occurrenceof acute respiratoryinfections in the first and second year of life, at least 12 months before the onset of disease, was associated to increased odds (> x2) of developing CD. It is most likely that viral infections (as the large majority of URTI in children) play a role in the development of food antigen intolerance leading to CD . A role of non-pathogenic viral infections has been also suggestedin the developmentof intolerance to gluten.
* No influence of breast-feeding or gluten introduction: breast feeding does not prevent the incidence of CD in at risk infants: its most likely effect is to delay the onset of clinical symptoms. Similarly, the time and quantity of gluten introduction is not associated to the actual incidence, but is only associated to delayed time effects.
* Possible implication of microbiome: despite the complexity of estimating differences in the composition of microbiome in the infants, it has been suggested that infants who later develop CD might show a fila composition slightly different from their matched controls.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women from a family with a confirmed CD proband

Exclusion Criteria:

Women affected by severe chronic disease and cancer Women not able to attend the schedule of visits

-

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women from a family with a confirmed CD proband Live newborns from the above mothers
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Celiac Disease | 6 years
  Number of new cases of infants affected by Celiac Disease in relation to genetic (HLA and non-HLA Associated Genes), Epigenetic (DNA Methylation, Gene Expression, Istone Acetylation of candidate gene) and environmental factors (Maternal factors, Nutrition, Infections)

SECONDARY OUTCOMES:
Analysis of microbiome | 6 years
  Difference in the microbiome composition of the group of infants who eventually develop Celiac Disease versus those who do not develop the disease.
  Comparison of Fecal Microbiome of infants at 4, 12 and 24 months subgrouped by outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Naples Azienda Ospedaliera Universitaria, Naples, Campania, Italy